CLINICAL TRIAL: NCT03475199
Title: Evaluation of FabLife's Personalised Support Program Effectiveness in Sperm Quality Improvement in Men Suffering From Hypofertility
Brief Title: Evaluation of Personalised Support Program Effectiveness in Sperm Quality Improvement
Acronym: FabLife
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FabLife (Industry)
Collaborators: Keyrus Biopharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-AO3218-45
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, controlled, national study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FabLife group (Experimental): Fablife personnalised support and telephone follow-up with a dietician.
  Interventions: Device: FabLife
- Control group (No Intervention): General dietary recommendations.

INTERVENTIONS:
Device: FabLife — * A personnalized dietary program depending on the patient's phenotype and genotype
  * The daily intake of a dietary supplement, developped in the context of male infertility.
  Arms: FabLife group

SUMMARY:
FabLife is an interventional, prospective, multicentre, controlled study undertaken in metropolitan France.

The main objective is to evaluate the effect of FabLife personalised program over a period of 15 weeks on the improvement of spermatic DNA fragmentation in subfertile men compared to general dietary recommendations.

DETAILED DESCRIPTION:
More than 15 % of couples couldn't get pregnant after at least a year of unprotected intercourse.

The FabLife personalised program aims to improve sperm quality including sperm DNA fragmentation in subfertile men through:

* A personalized dietary program based on patient's phenotype and genotype
* A daily dietary supplement, developed in the context of male infertility

A total of 75 patients will be recruited:

* 46 patients will benefit from the program,
* 23 patients will form the control group.
* 6 patients will not answer to all the criteria.

ELIGIBILITY:
Inclusion Criteria:

* All male volunteers aged 18 to 45 years belonging to a couple reporting an involuntary infertility greater than 12 months
* Conventional spermatic parameters compatible with spontaneous pregnancy

  * Sperm Count> 5M / ml and
  * Progressive sperm mobility> 20%
* Negative spermoculture
* Fragmentation of sperm DNA> 20%
* Patient able to understand dietary recommendations given in French, in writing and orally
* Social insured patient receiving benefits from the French Social Security health branch
* Patient with a mobile phone (iOS or Android) with internet access

Exclusion Criteria:

* Patient diagnosed with severe oligospermia (<5 million spz / ejaculate)
* Patient with BMI> 35 or <18.5
* Patient with known and treated diabetes
* Patient with known and treated lipid disorders
* Patient with known and treated cardiovascular diseases
* Patients with known and treated hypertension
* Patients with known and treated dysthyroidism
* Patients with known symptomatic varicocele
* Patient with known inflammatory bowel diseases
* Patient with renal failure diagnosed
* Patient presenting a viral risk (HIV / Hepatitis B and C / ...) requiring support in a dedicated circuit
* Patient unable to give informed consent
* Minors and protected adults, vulnerable people
* Patient participating in another clinical research study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Sperm DNA fragmentation | 15 weeks
  Difference in sperm DNA fragmentation from baseline to post-treatment

SECONDARY OUTCOMES:
Semen quality | 15 weeks
  Difference in semen quality (semen variables including total sperm count, sperm concentration, sperm motility, sperm morphology and semen volume) from baseline to post-treatment.
Sperm motility | 15 weeks
  Difference in sperm motility from baseline to post-treatment.
Sperm morphology | 15 weeks
  Difference in sperm morphology from baseline to post-treatment.
Sperm concentration | 15 weeks
  Difference in sperm concentration from baseline to post-treatment.
Semen volume | 15 weeks
  Difference in semen volume from baseline to post-treatment.
Total sperm count | 15 weeks
  Difference in total sperm count from baseline to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Levy, Md, PhD, Pr, Principal Investigator — Hopital Tenon (AP-HP) France
Locations (2):
- France (2):
  - Drouot Laboratory, Paris
  - Tenon Hospital (AP-HP), Paris